CLINICAL TRIAL: NCT06845826
Title: Point-of-Care High-Sensitivity Troponin Testing in the Emergency Department to Assess Myocardial Infarction for Timely Discharge
Brief Title: Point-of-Care Troponin Testing in the Emergency Department
Acronym: CERMIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Jan Verbakel, Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S68277
Record Dates: First submitted 2025-02-12; First posted 2025-02-25 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-02

CONDITIONS: Acute Coronary Syndromes
Keywords: POCT; troponine testing; acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: prospective, cross-sectional, interventional, single-center, open label, randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Usual care (No Intervention): care as usual: central laboratory troponine testing
- Intervention (Active Comparator): To establish in a randomized interventional controlled trial whether a novel POC test-guided strategy in acute chest pain patients in the ED results in a reduced length of stay compared to the usual central laboratory testing strategy when managing patients with a suspicion of NSTEMI
  Interventions: Device: Point-of-Care high-sensitivity troponin testing

INTERVENTIONS:
Device: Point-of-Care high-sensitivity troponin testing — To establish in a randomized interventional controlled trial whether a novel POC test-guided strategy in acute chest pain patients in the ED results in a reduced length of stay compared to the usual central laboratory testing strategy when managing patients with a suspicion of NSTEMI
  Arms: Intervention

SUMMARY:
The goal of this study is to evaluate whether a POC-guided testing strategy to exclude non-ST elevation myocardial infarction (NSTEMI) in acute chest pain patients presenting at the emergency department (ED) can result in a shorter length of stay compared to the routine central laboratory testing strategy. Currently, most often two high-sensitivity troponin (hs-cTn) tests are required for exclusion of NSTEMI, and central laboratories are struggling to achieve the recommended turnaround time of 60 minutes. Novel POC hs-cTn testing technology can provide results in minutes, potentially reducing the ED length of stay. This may lead to a reduction in ED crowding, which is a growing worldwide healthcare problem, resulting in poorer patient outcomes. This study may therefore improve patient burden, ED staff workload, and lead to more efficient expenditure of healthcare resources.

We will perform a prospective, cross-sectional, interventional, single-center, open label, randomized trial.

All consecutive patients older than 18 years and younger than 75 years presenting at the UZ Leuven emergency department with chest pain or chest pain-equivalent symptoms suspected of an acute coronary syndrome (ACS) will be invited to participate in the study. After informed consent patients will be randomized into the point-of-care testing (POCT) group or the usual care group. Patients in the POCT group will undergo the novel POC test-guided strategy. In the POC strategy the first hs-cTnI test shortly after admission to the ED will be performed on the POC Atellica VTLi. The second test will be performed with the usual central laboratory hs-cTnT test. Patients in the usual care group will undergo the usual testing strategy with one or two hs-cTnT tests performed in the hospital's central laboratory.

DETAILED DESCRIPTION:
Testing strategy Triage nurses, ED registration staff, or the treating physicians will identify eligible patients after which recruitment will be performed by the study collaborator(s). After informed consent patients will be randomized into the point-of-care testing (POCT) group or the usual care group. All patients first undergo usual work-up, including clinical history and examination, and an ECG, thereby identifying clinically unstable patients and patients with signs of a STEMI (exclusion criteria), and identifying patients who need further exclusion of a NSTEMI by hs-cTn testing. Patients in the POCT group will undergo the POC test-guided strategy with the Atellica VTLi. In the POC strategy the first hs-cTnI test shortly after admission to the ED will be performed on the POC Atellica VTLi. This represents a novel testing strategy. The second test will be performed with the usual central laboratory hs-cTnT test. Patients in the usual care group will undergo the traditional central laboratory hs-cTnT testing strategy. As a safety back-up in all patients in the POCT group, usual central laboratory high-sensitivity troponin testing will be performed as well. Only one additional blood sample tube is required to perform the POC test. The test requires a whole blood or plasma sample of 30-100 μL, which will be collected in a lithium-heparin tube. The sample can be safely transferred from the blood tube to the test cartridge with an accompanying transfer device designed by Siemens Healthineers at the point of care. The left-over material of the blood sample after POC testing will be transferred to the hospital's central laboratory to assess for the presence of haemolysis and its impact on the POC test results.

Management and treatment decisions The troponin test results will be available to the treating ED physicians, immediately influencing medical management decisions. The physicians will be trained correctly to use the POC device within the POC test-guided strategy. The Atellica VTLi will be connected to the laboratory information management system so the test result will be available in the patient's electronic medical health record (KWS). Patients in the POCT group presenting with chest pain after more than 3 hours of onset of the current episode of symptoms, no signs of ischaemia on ECG and with an hs-cTnI value below 7 ng/L on the Atellica VTLi will be considered at very-low risk for NSTEMI and can be considered for early ED discharge.(22) Patients with an hs-cTnI value higher than 60 ng/L are considered at high risk for NSTEMI and should be considered for immediate hospital admission and further treatment. Patients with an hs-cTnI value between 7 ng/L and 60 ng/L are considered at intermediate risk of NSTEMI and should be considered for a second hs-cTnT test within the standard UZ Leuven protocol. As a back-up in all patients in the POCT group an additional central laboratory hs-cTnT test will be performed, as POC test failures are currently seen in 7% of performed test, and since the test at admission is required to calculate the one-hour delta. The treating physician will be blinded to this test result to avoid waiting for a second confirmation of the POCT result and thereby compromising the ED length of stay. The result however will be communicated by the clinical laboratory to the treating physician in case of marked discrepant test results: if the result on the POC test is below 7 ng/L, allowing for rule-out of NSTEMI, while the result on the central laboratory test is > 14 ng/L, indicating a higher probability of NSTEMI. If the patient has already been discharged by the time the back-up test is communicated to the treating physician, the patient will be contacted to return to the ED for further examinations and further treatment if necessary. Re-admitted patients will be managed according to routine clinical care, and no additional study-related interventions will be applied. In the case of a negative POC test result, and a central lab hs-cTnT value between 5 and 14 ng/L, we deem the probability of an NSTEMI very low, allowing for ED discharge without further treatment. In case of a second test after 1 hour, the 0h hs-cTnT and the 1h hs-cTnT test will be reported together as usual through the electronic medical record, to allow for the assessment of a change in troponin values.

All final medical management decisions are at the discretion of the treating physician, so he or she is allowed to deviate from the proposed algorithm according to their clinical judgement. Other life-threatening causes of chest pain such as pulmonary embolisms, heart failure or pneumonia may be considered next to ACS. If the treating physician deems that NSTEMI is not sufficiently ruled out after a negative POC hs-cTnI test or other conditions should be further excluded, he or she is free to perform additional investigations or to admit the patient to a hospital ward. Patients in the usual care group will undergo usual central laboratory hs-cTnT testing.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures - At least 18 years of age at the time of signing the Informed Consent Form (ICF)
* Age < 75 years of age
* Presenting with chest pain or chest pain-equivalent symptom suspect of acute coronary syndrome at the University Hospitals Leuven emergency department; Symptoms must have (had) a minimum duration of 15 minutes, and the current, ongoing episode of symptoms must have started within the past 12 hours.

Exclusion Criteria:

* Unable to provide written informed consent
* Age <18 years or >75 years
* Chest pain or equivalent symptom with a duration shorter than 15 minutes, or an onset of the current, ongoing episode of symptoms more than 12 hours ago
* Clinically unstable patients or confirmed STEMI patients, requiring immediate treatment
* Patients with recent chest trauma
* Patients transferred from another hospital
* Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the CISP.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1552 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Length of stay at emergency department | Hours: 24
  with a tracking bracelet we measure the time of presentation until discharge of the patient in the emergency department

SECONDARY OUTCOMES:
30-day MACE | Day: 30
  To assess the secondary endpoint of major adverse cardiac events (MACE), the final diagnosis after the ED visit will be extracted from the electronic hospital patient record. For patients discharged home from the ED, thirty days after discharge the patient's hospital record will be checked and the patient's regular GP will be contacted to confirm if any major adverse cardiac events occurred.

OTHER OUTCOMES:
Degree of user friendliness: questionnaires and qualitative think aloud sessions | Hours: 24
  user friendliness of the POC Atellica VTLi hs-cTnI test device: questionnaires and think aloud sessions for qualitative research
Phyisican adherence | Hours: 24
  The physician will be asked to indicate whether the proposed testing strategy was followed or whether he or she deviated from it and the reason why, to assess the physician adherence to the testing strategy.
Patient satisfaction | Day: 7
  Patient satisfaction with the POC test-guided strategy will be assessed as an exploratory endpoint by contacting the patients after discharge (at day 7 baseline visit) and taking questionnaires on how they experienced their care. The Short Assessment of Patient Satisfaction (SAPS-)questionnaire will be used, extended with open questions and specific questions to our current study. Scoring is done by first reversing the scores for items #1, #3, #5, #7, and then summing all scores.
  The score range is from 0 (extremely dissatisfied) to 28 (extremely satisfied)
Comparison of POC and central laboratory hs-cTnI testing, and central laboratory hs-cTnT testing | Hours: 24
  Congruence between POC and central laboratory hs-cTnI testing, and central laboratory hs-cTnT testing: assessment of agreement in terms of diagnostic accuracy and correlation
External validation of clinical prediction models Heart score + T-MACS score | after obtaining the sample size
  Discrimination (AUC, O:E ratio, sensitivity and specificity), calibration and clinical utility (net benefit) of Heart score + T-MACS score

CONTACTS AND LOCATIONS:
Overall Officials: Jan YJ Verbakel, MD, PhD, Professor, Study Director — Leuven Unit for Health Technology Assessment Research, University of Leuven
Locations (1):
- KU/ UZ Leuven ED, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided